CLINICAL TRIAL: NCT00766493
Title: GORE® Embolic Filter in Carotid Stenting for High Risk Surgical Subjects (GORE EMBOLDEN)
Brief Title: GORE® Embolic Filter in Carotid Stenting for High Risk Surgical Subjects (EMBOLDEN)
Acronym: EMBOLDEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEF-06-08
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stenosis; embolic protection device; distal embolic filter; minimizing risks of carotid artery stenting
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GORE® Embolic Filter (Experimental): Subjects treated with the GORE® Embolic Filter and an FDA-approved carotid stent.
  Interventions: Device: GORE® Embolic Filter

INTERVENTIONS:
Device: GORE® Embolic Filter — Embolic protection during carotid stenting

SUMMARY:
Compare the 30-day safety and efficacy of the GORE® Embolic Filter used in conjunction with FDA-approved carotid stents to a performance goal obtained from carotid stent studies utilizing distal embolic protection.

DETAILED DESCRIPTION:
Continuous advances in angioplasty techniques and the development of low-profile, flexible, tapered nitinol stents designed specifically for carotid applications have made CAS a viable alternative to CEA. Advances in embolic protection technology will assist in moving CAS forward as a universally accepted procedure. While the GORE® Embolic Filter is similar in many ways to other currently available filters, it has been designed to provide optimal vessel wall apposition. Bench tests suggest that the wall apposition may provide improved filter efficiency, thereby minimizing embolization of particles downstream and potentially decreasing adverse clinical effects. In addition, preclinical testing suggests that the GORE® Embolic Filter has improved deliverability, including torque ability and lesion cross that may improve the ability of the system to access and treat tight lesions in tortuous anatomy. Thus, the purpose of this multi-center clinical study is to assess the safety and effectiveness of the GORE® Embolic Filter when used to provide cerebral embolic protection during carotid artery angioplasty and stenting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is either:

   * Symptomatic (amaurosis fugax in the hemisphere supplied by the target vessel, TIA or non-disabling stroke within 6 months of the procedure) with carotid stenosis ≥50% as diagnosed by angiography using NASCET methodology, OR
   * Asymptomatic with carotid stenosis ≥80% as diagnosed by angiography using NASCET methodology
2. Target lesion is located in one of the following:

   * ICA
   * bifurcation
   * CCA proximal to the bifurcation
3. At Anatomic risk for adverse events from CEA (e.g., restenosis after a prior CEA) or at Co-morbid risk for adverse events from CEA (e.g., unstable angina with ECG changes)

Exclusion Criteria:

* Recent surgical procedure within 30 days before or after the stent procedure
* Uncontrolled sensitivity to contrast media
* Renal Insufficiency
* Recent evolving, acute stroke within 21 days of study evaluation
* Myocardial infarction within 72 hours prior to stent procedure
* History of a prior major ipsilateral stroke with residual neurological deficits likely to confound the neurological assessments (e.g., NIHSS)
* Neurological deficits not due to stroke likely to confound the neurological assessments (e.g., NIHSS)

Angiographic Exclusion Criteria:

* Isolated ipsilateral hemisphere leading to subject intolerance to reverse flow
* Total occlusion of the ipsilateral carotid artery
* Pre-existing stent in the ipsilateral carotid artery OR the contralateral carotid artery that extends into the aortic arch
* Presence of a filling defect, thrombus, occlusion or "string sign" in the target vessel
* Severe lesion calcification restricting stent deployment
* Carotid stenosis located distal to target stenosis that is more severe than target stenosis
* >50% stenosis of the CCA proximal to target vessel
* Known mobile plaque in the aortic arch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A. Gray, MD, Principal Investigator — Columbia University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study will be conducted at a maximum of 40 medical institutions in the United States (including public and academic research center hospitals and private practices) and will enroll approximately 250 subjects.
Groups:
- EMBOLDEN: GORE® Embolic Filter with carotid artery stenting
Period: Pre-Discharge
Arm/Group | EMBOLDEN
Started | 250
Completed | 250
Not Completed | 0
Period: 30 Days Post-Procedure
Arm/Group | EMBOLDEN
Started | 250
Completed | 238
Not Completed | 12
Not completed — Discontinued | 7
Not completed — Missed Visit - Phone Contact f/u | 4
Not completed — Missed Visit - No Phone Contact | 1

BASELINE CHARACTERISTICS:
Arm/Group | EMBOLDEN
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (9.4)
Age, Continuous [Median (Full Range); unit: Years] | 74.7 [51.3 to 92.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 153
History of Diabetes [Number; unit: Participants]
  Yes | 87
  No | 163
History of Hypertension [Number; unit: Participants]
  Yes | 236
  No | 14
History of Ischemic Stroke [Number; unit: Participants]
  None | 200
  One | 34
  Two or More | 12
  Unknown | 4
Previous Endarterectomy [Number; unit: Participants]
  None | 171
  Less than 1 Year | 13
  1 Year or Greater | 63
  Unknown | 3
Symptomatology [Number; unit: Participants]
  Symptomatic | 37
  Asymptomatic | 213

OUTCOME MEASURES:

1. Primary Outcome: Composite Major Adverse Event (MAE) Rate of Death, Myocardial Infarction, and Stroke at 30 Days Postprocedure
Time Frame: 30 days
Population: EMBOLDEN subjects evaluable for the primary endpoint
Measure: Number; unit: Participants
Arm/Group | EMBOLDEN
Number analyzed (Participants) | 234
Participants
  Subjects With One or More Major Adverse Events | 10
  Death | 2
  Myocardial Infarction (MI - Overall) | 1
  Q-Wave MI | 0
  Non-Q-Wave MI | 1
  Stroke (Overall) | 7
  Major Stroke (Overall) | 1
  Ischemic Stroke (Major) | 1
  Hemorrhagic Stroke (Major) | 0
  Minor Stroke (Overall) | 6
  Ischemic Stroke (Minor) | 6
  Hemorrhagic Stroke (Minor) | 0
Statistical Analysis 1: Comparison: EMBOLDEN; This study is designed to test the primary null hypothesis that the composite MAE outcome of all death, stroke, and/or MI when using the GORE Embolic Filter is equal to or higher than a Performance Goal (PG) of 6.4% established from published carotid stenting studies utilizing distal embolic protection, versus the alternative hypothesis that the composite MAE outcome is less than the performance goal. The sample size was calculated based on 80% power and a 1-sided Type I error rate of 0.025; Test type: Superiority or Other; p = 0.0001, One Sample Binomial — Reject H0 if z<-1.96, or 1-sided p<0.025; Significance test was based on a one-sample normal approximation to the binomial test; Proportion = 0.043, 95% CI 2-sided [0.021 to 0.077], Standard Error of Mean 0.013 — The 2-sided 95% CI is reported for descriptive purposes; the statistical hypothesis test is 1-sided

2. Secondary Outcome: Device Success
Description: Device Success defined as the number of participants with Technical Success using the GORE Embolic Protection System (i.e., the GORE Embolic Filter device was delivered, placed, and retrieved as outlined in the Instructions for Use).
Time Frame: Post Procedure
Measure: Number; unit: Participants
Arm/Group | EMBOLDEN
Number analyzed (Participants) | 250
Participants | 241

3. Secondary Outcome: Clinical Success
Description: Clinical Success defined as GORE Embolic Filter and carotid stent success in the absence of death, emergency endarterectomy, repeat PTA / thrombolysis of the target vessel, and stroke or MI as determined by the Clinical Events Committee. Clinical success will be evaluated from procedure through 24-48 hours postprocedure.
Time Frame: 30 days
Measure: Number; unit: Participants
Arm/Group | EMBOLDEN
Number analyzed (Participants) | 250
Participants | 233

4. Secondary Outcome: Access Site Complications
Description: Access Site Complications defined as the presence of a large hematoma (>5cm or requiring treatment or prolonged hospitalization), fistula or pseudoaneurysm formation, retroperitoneal bleeding or the need for surgical repair postprocedure.
Time Frame: 30 days
Measure: Number; unit: Participants
Arm/Group | EMBOLDEN
Number analyzed (Participants) | 250
Participants | 6

5. Secondary Outcome: Neurologic Events
Description: Neurological Events at 30 days post-procedure, including transient ischemic attacks (TIAs).
Time Frame: 30 days
Measure: Number; unit: Participants
Arm/Group | EMBOLDEN
Number analyzed (Participants) | 250
Participants | 16

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | EMBOLDEN
Serious Adverse Events (participants affected / at risk) | 56/250
Other Adverse Events (participants affected / at risk) | 83/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMBOLDEN (N=250)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Blood & Lymphatic System - Other (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 5 (5)
Angina/coronary ischemia (Cardiac disorders) | 3 (3)
Asystole (Cardiac disorders) | 2 (2)
Cardiac - Other (Cardiac disorders) | 3 (3)
Congestive Heart Failure (CHF) - onset or worsening of (Cardiac disorders) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (MI) (Cardiac disorders) | 1 (1)
Thrombosis/Occlusion - GEF (Surgical and medical procedures) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1)
Retroperitoneal bleed (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Groin Hematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3)
Infection at access site (Injury, poisoning and procedural complications) | 1 (1)
Metabolism & Nutrition - Other (Metabolism and nutrition disorders) | 1 (2)
Musculoskeletal and Connective Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous System - Other (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Cerebral ischemia/transient ischemic attack (TIA) (Nervous system disorders) | 2 (2)
Visual disturbance (Nervous system disorders) | 1 (1)
Stroke/cerebrovascular accident (CVA) (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 2 (2)
Ischemic stroke (Nervous system disorders) | 1 (1)
Renal failure/insufficiency (Renal and urinary disorders) | 1 (1)
Renal & Urinary - Other (Renal and urinary disorders) | 2 (2)
Respiratory, Thoracic & Mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
COPD, worsening of (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 14 (14)
Hypertension (Vascular disorders) | 2 (2)
Bleeding (Vascular disorders) | 1 (1)
Vessel spasm (Vascular disorders) | 1 (1)
Vascular - Other (Vascular disorders) | 2 (2)
Ischemia/Infarction of tissue/organ (Vascular disorders) | 2 (2)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Vessel dissection, perforation or rupture (Vascular disorders) | 1 (1)
Not Elsewhere Classified - Other (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMBOLDEN (N=250)
Anemia (Blood and lymphatic system disorders) | 14 (14)
Bradycardia (Cardiac disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 12 (12)
Nervous System - Other (Nervous system disorders) | 14 (15)
Headache (Nervous system disorders) | 11 (11)
Hypotension (Vascular disorders) | 38 (39)
Hypertension (Vascular disorders) | 16 (16)
Bleeding (Vascular disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.